CLINICAL TRIAL: NCT02742532
Title: Oxytocin Suppresses Substance Use Disorders Associated With Chronic Stress
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jennifer Mitchell (Other)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); Congressionally Directed Medical Research Programs (U.S. Federal Agency); Eisenhower Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Jennifer Mitchell, Associate Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NMCSD Oxytocin
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Alcohol Use Disorder; Stress Disorders, Post-Traumatic; Anxiety Disorders; Substance Use Disorders
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic; Anxiety Disorders; Substance-Related Disorders | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): Intra-nasal oxytocin (40 IUs; 5 puffs in each nostril)
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Intra-nasal saline placebo (5 puffs in each nostril)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Intranasal oxytocin 40 IU
  Other Names: Syntocinon nasal spray
  Arms: Oxytocin
Drug: Placebo — Intranasal saline solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether oxytocin will decrease craving to use drugs/alcohol and stress reactivity following exposure to laboratory-induced stress among Active Duty Service Members with a dual diagnosis of alcohol/substance use disorder (ASUD) and post-traumatic anxiety.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether intra-nasally administered oxytocin will decrease craving to use alcohol and stress reactivity following exposure to laboratory-induced stress among Active Duty Service Members (AD SMs) with a dual diagnosis of alcohol/substance use disorder (ASUD) and post-traumatic anxiety (i.e., PTSD or anxiety disorder NOS).

This is a 2-arm placebo controlled study. Subjects will complete a battery of self-report questionnaires and behavioral interviews. Baseline assessments of subjective (craving, stress), physiologic (HR, BP), and neuroendocrine measures (salivary cortisol) will be collected. These same assessments will be repeatedly collected throughout the testing portion of the study. Subjects will receive acute administration of intra-nasal oxytocin or placebo and will then be exposed to a laboratory-induced social stressor. They will be asked to give a short speech and perform arithmetic in front of a panel of judges. Following the task, additional post-task assessments of the subjective, physiological, and neuroendocrine measures will be completed over the next hour.

ELIGIBILITY:
Inclusion Criteria:

* Active Duty Service Members, any service branch; age 18-65 years.
* Meets clinician assessment for current PTSD OR anxiety disorder NOS OR scores on DASS > 10 on Anxiety or > 19 on Stress.
* Meets clinician assessment for alcohol use disorder (AUD) OR scores >8 on AUDIT.
* If meet current or lifetime criteria for another substance disorder, must indicate that AUD is primary.
* Subjects taking psychotropic medications will be required to be maintained on a stable dose for at least two weeks before study initiation (unless at physician's discretion following psychological consult).
* Negative urine drug screen test and BAC =0.
* Able to comprehend English.
* Able to provide informed consent and function at an intellectual level sufficient to allow completion of the assessment instruments.
* Must consent to random assignment to oxytocin or placebo.

Exclusion Criteria:

* Positive urine drug screen (except marijuana) or BAC > 0.
* Untreated subjects currently symptomatic of psychotic or bipolar affective disorders.
* Subjects with current suicidal or homicidal ideation and intent, who would present a serious suicide risk.
* Subjects on psychotropic drugs that have been initiated during the past 2 weeks (unless approved at physician's discretion following psychological consult).
* Subjects with a history of a major medical illness (e.g., endocrine, cardiovascular, central nervous system disorders, peripheral neuropathy, or pulmonary disease) or other acute or unstable medical condition that might interfere with safe conduct of the study or accurate interpretation of the results.
* Subjects experiencing withdrawal symptoms as reported by Clinician or systolic BP≥160 mmHg, diastolic BP ≥100 mmHg and resting HR ≥100 bpm.
* Subject is considered unsuitable for the study in the opinion of study PI or AIs for any other reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mardi Smith, PhD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin | Placebo
Started | 31 | 32
Completed | 28 | 31
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 32 | 63
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 27.09 [19 to 45] | 27.38 [20 to 42] | 27.24 [19 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 26 | 29 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 2 | 0 | 2
  White | 25 | 29 | 54
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 32 | 63
Self-Reported Alcoholic drinks per week [Mean (Standard Deviation); unit: standard drinks/week] — Population: Some subjects declined to complete this data, so the row population differs from the overall.
  standard drinks/week
    number analyzed (Participants) | 28 | 30 | 58
    (all) | 51.2 (39.9) | 43.9 (45.9) | 47.4 (42.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Craving to Use Alcohol Rating (Visual Analog Scale)
Description: The Visual Analog Scale (VAS) is a horizontal line of fixed 100 mm length. The ends are defined as the extreme limits of the parameter from the left (least) to the right (most). Subjects mark the point on the line that represents their perception of the parameter. The score is determined by measuring in millimeters from the left end of the line to the point that the patient marks. The score range is 0-100, with higher scores indicating higher cravings.
Time Frame: Change from baseline to post-drug at 20 minutes
Population: All subjects who completed this outcome measure were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 29 | 32
score on a scale | 0.076 (1.77) | -0.928 (1.42)

2. Secondary Outcome: Change in Stress Rating (Visual Analog Scale)
Description: The Visual Analog Scale (VAS) is a horizontal line of fixed 100 mm length. The ends are defined as the extreme limits of the parameter from the left (least) to the right (most). Subjects mark the point on the line that represents their perception of the parameter. The score is determined by measuring in millimeters from the left end of the line to the point that the patient marks. The score range is 0-100, with higher scores indicating higher stress.
Time Frame: Change from baseline to post-drug at 20 minutes
Population: All subjects who completed this outcome measure were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 29 | 32
score on a scale | -0.755 (1.24) | -1.268 (1.82)

ADVERSE EVENTS:
Time Frame: From enrollment through study completion, an average of 1 year
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 0/31 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT02742532/Prot_SAP_001.pdf